CLINICAL TRIAL: NCT06243276
Title: Effects of Diabetes on Two Short Implants Splinted Using One- and Two-stage Techniques: Split-mouth Study With One-year Follow-up.
Brief Title: Effect of Diabetes on Short İmplants in One- and Two-Stage Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan University (Other)
Collaborators: Mode Medical Implant Manufacturer (Unknown)
Responsible Party: Principal Investigator, Ömer Faruk Okumuş, Assistant Professor, Erzincan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EUDF-OKUMUS-002
Record Dates: First submitted 2024-01-18; First posted 2024-02-06 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Dental Implant Surgical Techniques; Diabetes Mellitus; Short Dental Implants
Keywords: Dental Implants; Short Dental Implants; One Stage Implant Surgery; Two Stage Implant Surgery; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Split-mouth study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic patients (Active Comparator)
  Interventions: Procedure: One stage implant surgery; Procedure: Two stage implant surgery
- Healthy patient (Active Comparator)
  Interventions: Procedure: One stage implant surgery; Procedure: Two stage implant surgery

INTERVENTIONS:
Procedure: One stage implant surgery — It is a technique in which the healing cap is connected to the implant at the stage of implant placement.
Procedure: Two stage implant surgery — It is a technique in which the healing cap is connected to the implant three months after the implant is placed.

SUMMARY:
The goal of this clinical trial is to compare one- and two-stage techniques for short implant surgery in diabetes. The main questions it aims to answer are:

* Is one-stage short implant surgery at risk of implant osseointegration in diabetic patients compared to two-stage surgery?
* Is one-stage short implant surgery associated with a risk of implant survival (at one-year follow-up) in diabetic patients compared to two-stage surgery?
* What are the effects of one- and two-stage short implant surgery on the marginal bone loss or ISQ (implant stability coefficient - resonance frequency analysis device measurement) values of the implant in diabetic patients?

Participants will come for their 3rd, 6th and 12th month controls.

* Participants will receive two adjacent short implants.
* A randomly selected one of these short implants will undergo a one-stage implant surgery, and the other a two-stage implant surgery.
* Data will be obtained through non-invasive evaluation methods during the surgery and subsequent control stages.

Researchers will also test one- and two-stage short implant surgeries in a control group of healthy individuals. Thus, the effects of diabetes on these two techniques will be better understood by comparing them with the healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* The maxillary and mandibular posterior region (distal part of the canine in each quadrant) must have toothless space for two adjacent short implants.
* The edentulous space must have a vertical bone height of at least 5 mm. (Distance to maxillary sinus and alveolar nerve)
* The edentulous space should not require horizontal bone augmentation. (for implants with diameters 3.7 - 4.1 - 4.7 - 5.3)
* Bleeding on probing should be less than 10%. There should be no pathological pockets in any tooth.
* Participant should not smoke more than 10 cigarettes per day.
* More than 6 months must have passed since the tooth extraction from the edentulous area.
* Should not have bruxism
* If it is diabetes, the HbA1c value should be greater than 6.5, and if it is healthy control, the HbA1c value should be between 4 and 5.

Exclusion Criteria:

* Having psychological problems
* Smoking more than 10 cigarettes per day
* Pregnancy status if female patient
* Having a medication or disease that will cause abnormal post-operative bleeding
* Alcohol and drug use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06-05 (Estimated); Primary Completion 2024-06-14 (Estimated); Study Completion 2025-05-14 (Estimated)

PRIMARY OUTCOMES:
One-year survival of the implant | At the end of 12 months of follow-up from the surgery in which the implant was placed in the bone
  To observe whether the implant is performing its function. The implant continues to support the tooth connected to it.
Evaluation of the status of osseointegration | Three months after the implant is placed in the bone. (At the end of three months)
  Fusion of the dental implant with the bone at the microscopic level. Osseointegration will be evaluated as successful or unsuccessful. Successful osseointegration is defined by no mobility in the implant, no radiolucency around the implant on radiography, and no pain in the implant. Otherwise, the osseointegration of the implant is considered unsuccessful.

SECONDARY OUTCOMES:
Implant Stability Quotient (ISQ Value) | 1- Surgical stage where the implant is placed; 2- Three months after the implant is placed in the bone. At the end of three months
  The value obtained by the resonance frequency analysis (RFA) device used to measure the primary stability of dental implants. The RFA technique is based on continual excitation of the implant through dynamic vibration analysis. A transducer is connected to an implant, which is excited over a range of sound frequencies with subsequent measurement of the vibratory oscillation of the implant. It is a non-invasive technique.
Marginal bone level change | 1- Surgical stage where the implant is placed; 2- Three months after the implant is placed in the bone; 3- Six months after the implant is placed in the bone; 4- Twelve months after the implant is placed in the bone
  It defines the change in the marginal bone level in the neck area of the implant. It is determined by radiographic examination. The initial radiograph is compared with the radiograph at the end of three months. In measurements where the implant platform is the reference point, bone level changes are calculated in mm.